CLINICAL TRIAL: NCT07375043
Title: Drumming Groups for Parents of Autistic Children
Acronym: DG_PAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Eugenia Hernandez-Ruiz, Associate Professor of Music Therapy, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00022914
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Acute; Stress; Depression and Quality of Life; Stress in Parents of Autistic Children
Keywords: autism; stress; parents; caregivers; anxiety; depression
MeSH Terms: conditions — Depression; Autistic Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Parents will participate in drumming sessions that teach stress management techniques, sense of belonging, and coping skills for depression and anxiety.
  Interventions: Behavioral: Group Drumming

INTERVENTIONS:
Behavioral: Group Drumming — This Drumming program is based on HealthRhythms®, a drumming protocol that has been used extensively in clinical and community populations and has research support (e.g., Grab et al., 2023; Stevens & Fowl, 2024; Wachi et al., 2007). Adaptations will be derived from the PI's clinical and research experience with parents of autistic children. Each drumming session will have the following structure: introduction to the program, light movement & music, icebreakers with small percussions, technique pointers for percussion instruments, rhythmic introductions (sharing names with a percussive rhythm), free group drumming, soundscapes (creating visualizations with drumming), verbal processing, closing drumming exercise. The soundscapes are creative outlets to "paint a picture" with music. These exercises promote community, engagement, emotional expression, and creative thinking, which reduce stress. Specific strategies will include reflecting, mirroring, validating, and solution reframing.

SUMMARY:
This project aims to encourage a sense of belonging, community, and emotional support for parents of autistic children through a group drumming (music therapy) intervention.

DETAILED DESCRIPTION:
This pilot one-group pretest-posttest study will investigate the limited efficacy and acceptability of an 8-week drumming group on immediate stress (pre-post session) as measured by the STAI-S Short Form scale (Spielberger, 1977); on anxiety and depressive symptoms, as measured by the K-10 scale (Kessler et al., 2002) before and after the 8-week program, and group cohesion and acceptability as measured by the Group Therapy Experience Scale (GTES, Marziliano et al., 2018) after the program. As a group setting, this program does not substitute clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* parents or main caregivers of children in the Autism Spectrum,
* able to read and write in English.
* 18 years or older

Exclusion Criteria:

* Paid caregivers
* Unable to speak, read and write in English
* Unable to follow instructions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
K-10 | Pretest at the beginning of the first weekly session, and posttest at the end of the 8th weekly session.
  Anxiety and depressive symptoms, as measured by the K-10 scale (Kessler et al., 2002). Maximum score is 50, with each of the 10 items scored 1 to 5. Higher scores indicate higher distress. Optimal cutoff scores for clinically significant nonspecific psychological distress and need for treatment: total score =12, Depression = 7, and Anxiety = 3/4 (Lace et al., 2019).
STAI-S | Pretest at the beginning of the first weekly session, and posttest at the end of the 8th weekly session.
  Measures of state anxiety as measured by the State Trait Anxiety Inventory for Adults- Short Form Y1 (STAIAD-S Y1) scale (Spielberger, 1977). Maximum score is 40, with each of the 10 items scored 1 to 4, and four reverse-coded items. Higher scores indicate less anxiety (more wellbeing).
GTES | Posttest at the end of the 8th weekly session.
  Group cohesion and acceptability as measured by the Group Therapy Experience Scale (GTES, Marziliano et al., 2018). Maximum score is 80 with each of the 16 items scored from 1 to 5. Higher scores indicate better group experience.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Hernandez Ruiz, PhD, Principal Investigator — Arizona State University
Locations (1):
- Gateway Building, Room 361 & 363, Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will make the data available upon written request
Supporting Information: Study Protocol, CSR
Time Frame: January 2027 -December 2031
Access Criteria: Investigators with a minimum of a PhD education and institutional affiliation may request aggregated, anonymized data. Raw, anonymized data would be available to researchers in reputable research organizations if an approved study protocol for secondary data analysis is shared with the PI.
URL: https://search.asu.edu/profile/3309676